CLINICAL TRIAL: NCT06004908
Title: Role of MRI in Diagnosis of Causes of Postmenopausal Bleeding in Correlation to Histopathological Results
Brief Title: Role of MRI in Diagnosis of Postmenopausal Bleeding Causes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kholoud Khaled Salem Ali, Assistant lecturer, Assiut University
Other Study IDs: MR imaging in uterus
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Postmenopausal Bleeding
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — a type of scan that uses strong magnetic field sand radio waves to produce detailed images of the inside of the body
  Other Names: Magnetic resonance imaging

SUMMARY:
The aim of the study is to determine the diagnostic performance of MRI of endometrial pathology in postmenopausal women with postmenopausal bleeding

DETAILED DESCRIPTION:
Postmenopausal bleeding is a common clinical problem accounting for approximately 5% of office visits to a general gynecologist.

Postmenopausal bleeding has been defined as:

1. Vaginal bleeding occurring at least 6 months after complete cessation of menses in women not on hormonal replacement therapy (HRT).
2. Noncyclic vaginal bleeding occurring in postmenopausal women who are receiving HRT Abnormal vaginal bleeding may be caused by a number of gynecologic or nongynecologic disorders. When evaluating a gynecologic etiology, the primary goal is to eliminate the possibility of endometrial cancer which is the cause of bleeding in approximately 10% of postmenopausal women presenting with this complaint and is the presenting symptom in 90% of women with endometrial cancer.

Other common gynecologic etiologies include endometrial polyps, endometrial hyperplasia, and submucosal fibroids along with the use of hormone replacement therapy, tamoxifen, and phytoestrogens Those pathologies should be discriminated to navigate the treatment process. Transvaginal ultrasonography (TVS) is the most efficient first-step technique for diagnosis of postmenopausal bleeding . The sensitivity of TVS to detect endometrial pathologies is high, but its specificity is low . Therefore, biopsy is recommended as a second-step diagnostic method when endometrial thickness exceeds 4 mm . However, endometrial biopsy or dilatation and curettage (D&C) may not be possible in postmenopausal patients due to endometrial atrophy, endometrial adhesions, or the requirement of general anesthesia. . Furthermore, besides pain and discomfort with endometrial sampling procedures, in some occasions such as vaginal/cervical stenosis or pelvic organ prolapse these procedures may be difficult to be done . Additionally, blind sampling may not be an effective approach for diagnosis of focal endometrial lesions and may be subject to sampling error .

MRI is an emerging modality for various reasons, such as exquisite soft-tissue resolution, its capability of multiplanar imaging, characterization, high sensitivity, and lack of ionizing radiation.

The sensitivity of MRI in identifying acute uterine pathologies is 96.6 % With recent advances in MR imaging techniques, diffusion weighted (DW) imaging and ADC value are useful in characterization of endometrial lesions because malignant lesions show high cellularity with little extracellular space which give restricted motion of water molecules and lower ADC values in contrast to benign lesions and normal tissues .

ELIGIBILITY:
Inclusion Criteria:

1. Any female patient after menopause suffering from vaginal bleeding.
2. Patients receiving tamoxifen with vaginal bleeding.
3. Patient had histopathological biopsy examination either by total hysterectomy, hysteroscopy or D &C.
4. Patient must have local cause

   -

   Exclusion Criteria:

1. Patients not amenable for MRI examination 2. Patients not in menopause 3. Patients have general bleeding tendency 4. Patients not underwent histopathological biopsy examination

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any female patient after menopause suffering from vaginal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
comparison between pre-biopsy MRI based diagnosis and histopathological proved diagnosis in cases of post-menopausal vaginal bleeding | baseline
  anaylsis between pre-biopsy MRI based diagnosis and histopathological proved diagnosis in cases of post-menopausal vaginal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Hossam ElDen Mustafa Kamel, MD, Principal Investigator — unaffilitated

REFERENCES:
- [Background] Dubinsky TJ, Parvey HR, Maklad N. The role of transvaginal sonography and endometrial biopsy in the evaluation of peri- and postmenopausal bleeding. AJR Am J Roentgenol. 1997 Jul;169(1):145-9. doi: 10.2214/ajr.169.1.9207515.
- [Background] Karlsson B, Granberg S, Wikland M, Ylostalo P, Torvid K, Marsal K, Valentin L. Transvaginal ultrasonography of the endometrium in women with postmenopausal bleeding--a Nordic multicenter study. Am J Obstet Gynecol. 1995 May;172(5):1488-94. doi: 10.1016/0002-9378(95)90483-2. PMID 7755059
- [Background] Gull B, Karlsson B, Milsom I, Granberg S. Can ultrasound replace dilation and curettage? A longitudinal evaluation of postmenopausal bleeding and transvaginal sonographic measurement of the endometrium as predictors of endometrial cancer. Am J Obstet Gynecol. 2003 Feb;188(2):401-8. doi: 10.1067/mob.2003.154. PMID 12592247
- [Background] Foti PV, Tonolini M, Costanzo V, Mammino L, Palmucci S, Cianci A, Ettorre GC, Basile A. Cross-sectional imaging of acute gynaecologic disorders: CT and MRI findings with differential diagnosis-part II: uterine emergencies and pelvic inflammatory disease. Insights Imaging. 2019 Dec 20;10(1):118. doi: 10.1186/s13244-019-0807-6. PMID 31858287